CLINICAL TRIAL: NCT05154188
Title: Post Approval Study to Assure the ContInued saFety and effectIveness of Neuro Cochlear Implant System in Adult Users
Acronym: PACIFIC
Status: Not yet recruiting | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP25
Record Dates: First submitted 2021-10-13; First posted 2021-12-13 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Sensorineural Hearing Loss, Bilateral; Sensorineural Hearing Loss, Severe; Sensorineural Hearing Loss, Profound
Keywords: candidates for a cochlear implantation surgery; patients aged 18 years and older
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Neuro Cochlear Implant system — Patients will be regular candidates for a cochlear implantation surgery, according to the indication criteria of the Neuro Cochlear Implant System and the device will be used according to its intended purpose
  Other Names: Neuro ZtiCLA implant; Neuro ZtiEVO implant; Neuro 2 Sound Processor; Neuro 2 SP; Neuro Zti

SUMMARY:
On June 23, 2021, the Oticon Medical Neuro Cochlear Implant System (NCIS) was granted premarket approval (PMA) in the US to treat individuals 18 years or older, with bilateral severe-to-profound sensorineural hearing loss, who obtain limited benefit from appropriately fitted hearing aid(s).

To help assure the continued safety and effectiveness of an approved device, a post-approval study was required as a condition of approval under 21 CFR 814.82(a)(2).

The purpose of this study is to provide longer-term data on the safety and effectiveness of the Neuro Cochlear Implant System under general conditions of use in the postmarket environment.

DETAILED DESCRIPTION:
The post-approval study will be an open-label, prospective, multi-center, single-arm, non-randomized, self-controlled clinical trial in 10 clinical sites in the US.

The purpose of this study is to provide longer-term data on the safety and effectiveness of the Neuro Cochlear Implant System under general conditions of use in the postmarket environment. This study will be conducted as a prospective, non-controlled, non-randomized study in 10 clinical sites.

A total of 60 subjects, newly treated will be enrolled. Study subjects will be followed for 3 years post implantation of the device with a target follow-up rate of 80% at the end of the study

The primary safety endpoint is the comparison of the type and frequency of adverse events and serious adverse events observed during the study period. The effectiveness endpoints will include the within-subject differences for sentence recognition as evaluated with the AzBio test.

The study will include the following visits: baseline, 1-month post-surgery (activation date), 3 months, 6-months, 12-months, 18-months, 24-months, and 36-months post-activation. Each participant will serve as their own control with baseline measurements.

The total estimated duration of the study is 60 months: 24 months of recruitment and 36 months of subject participation.

The first patient is expected to be included within 6 months of study approval (obtained on August 19, 2021).

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age or older
* Obtain limited benefit from appropriately fitted hearing aids
* Bilateral severe-to-profound sensorineural hearing loss _ Severe-to-profound hearing loss is determined by a pure-tone average (PTA) superior or equal (≥) to 70 dB HL at 500, 1000 and 2000 Hz. Limited benefit from amplification is defined by scores of 50% or less on a validated sentence recognition test in quiet (AzBio sentences), in the best-aided listening condition _

Exclusion Criteria:

* Previous cochlear implantation
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array
* Active external or middle ear infections or tympanic membrane perforation in the ear to be implanted
* Presence of medical contraindications to middle-ear or inner-ear surgery or anesthesia as required
* Diagnosis of retro-cochlear pathology
* Diagnosis of auditory neuropathy
* Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and use of the prosthetic device
* Unwillingness or inability to comply with all investigational requirements
* Additional cognitive, medical, or social handicaps that would prevent completion of all study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * The current post-approval study concerning the NCIS will enroll a total of 60 subjects, newly treated. Patients will be regular candidates for a cochlear implantation surgery, according to the indication criteria of the Neuro Cochlear Implant System and the device will be used according to its intended purpose.
  * 60 subjects must meet the eligibility criteria
  * The patient can be an existing audiology patient of the CI clinic or can be referred from an outside hearing aid clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Stability of improvement of speech perception performance at 12- and 36-months post-activation with AzBio sentence scores. | At 12- and 36-months post-activation (visit 9 and visit 11)
  Average scores for AzBio sentence tests will be recorded in Quiet at 12- and 36-months post-activation and compared to pre-operative (baseline) measures.
  The AzBio sentence test is a validated sentence recognition test in quiet and has a score range of 0-100% with higher values indicating better scores.
Safety outcome | From Visit 1(8- 12 weeks pre-surgery) to Visit 12 (36 Months post-activation)
  Occurrence and severity of all adverse events and serious adverse events occuring during the study period. All device failures (internal and external parts) will be documented.

SECONDARY OUTCOMES:
Stability of improvement of speech perception performance at 12- and 36-months post-activation with CNC-words scores. | At 12- and 36-months post-activation (visit 9 & visit 12)
  Consonant-Nucleus-Consonant (CNC) scores will be recorded in Quiet at 12- and 36-months post-activation and compared to pre-operative (baseline) measures.
  The CNC word test has a score range of 0-100% with higher values indicating better scores.
Stability of outcomes over time using AzBio Sentence scores at 1 month in Quiet. | At 1 month post-activation (Visit 6)
  Scores for AzBio sentence tests will be recorded in Quiet at 1-month post-activation in quiet and compared to pre-operative (baseline) measures.
  The AzBio sentence test is a validated sentence recognition test in quiet and has a score range of 0-100% with higher values indicating better scores.
Stability of outcomes over time using AzBio sentences in Quiet and Noise at 3- ; 6- and 24-months post-activation | at 3 months(visit 7), 6 months (visit 9) and 24 months (visit 11)
  Average scores for AzBio sentence tests will be recorded in Quiet at 3- ; 6- and 24-months post-activation and compared to pre-operative (baseline) measures.
  The AzBio sentence test is a validated sentence recognition test and has a score range of 0-100% with higher values indicating better scores.
Stability of outcomes over time using CNC word scores at 3-, 6- and 24-months | At 3 months(visit 7), 6 months (visit 9) and 24 months (visit 11)
  Average scores for CNC word test will be recorded at 3-, 6- and 24 months post-activation and compared to pre-operative (baseline) measures.
  The Consonant-Nucleus-Consonant (CNC) word test has a score range of 0-100% with higher values indicating better scores.
Stability of outcomes over time for patients under a bimodal condition (i.e., patient wearing a contralateral hearing aid). | At 3-months post activation (visit 7) and 12 months (visit 9)
  Average scores for AzBio sentence tests will be recorded in Noise (at +10dB SNR), at 3- and 12-months post-activation and compared to pre-operative (baseline) measures.
  The AzBio sentence test is a validated sentence recognition test and has a score range of 0-100% with higher values indicating better scores.
Longitudinal measures of patient reported outcomes in a newly-implanted population | At 6-,12-,24- and 36 months post-activation (Visits 8,9,11,12)
  Patient reported outcome (PRO) measures including quality of life, listening effort and tinnitus at 6-,12-,24- and 36 months post-activation
Longitudinal measures of cognitive abilities in a newly implanted population | At 12-24 and 36 months post-activation (Visits 9,11,12)
  Scores on a cognitive assessment at 12-24 and 36 months post-activation
Longitudinal programming parameters (T- and C- levels) | At activation (Visit 5), then from 3 months post-activation (V7) throught study completion (an average of 3 years post activation)
  T and C levels collected at all intervals
Longitudinal device functionality measures (impedances) | At activation (Visit 5), then from 3 months post-activation (V7) throught study completion (an average of 3 years post activation)
  Electrode impedances collected at all intervals
Pedictors of outcomes: Electrode impedances collected at all intervals | At surgery visit (Visit 3 baseline visit) then from activation, 1-month post surgery( visit 5) throught study completion (an average of 3 years post activation)
  Electrode impedances collected at all intervals
Pedictors of outcomes: eCAP responses collected in the operating room | From activation (visit 5) throught study completion (an average of 3 years post activation)
  eCAP responses collected in the operating room
Proportion of major postsurgical complications and AEs over time | At surgery visit (i.e. visit 3, baseline visit, )
  Surgeon perception of handling of the Neuro Zti and electrode array as well as information related to surgical technique

IPD SHARING:
Plan to Share IPD: No